CLINICAL TRIAL: NCT00595868
Title: Efficacy of Varenicline in Ambivalent Smokers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Vermont Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, John Hughes, Professor, University of Vermont Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIR GA3051DO; IIR GA3051DO (Other Grant/Funding Number: Pfizer)
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Results first posted 2011-11-22 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-11

CONDITIONS: Tobacco Use Disorder; Tobacco Use Cessation; Nicotine Dependence
Keywords: Nicotine; Smoking; Smoking Cessation
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use Cessation; Smoking; Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Varenicline (Experimental)
  Interventions: Drug: Varenicline
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — 0.5 milligrams two times per day for 3 days, then 1.0 milligrams two times per day for an addition 11 days - 2 months
  Other Names: Chantix
  Arms: Varenicline
Drug: Placebo — same as Varenicline arm
  Arms: Placebo

SUMMARY:
The purpose of this study is to test whether Varenicline can help ambivalent smokers (those who are interested in quitting at some point in the future but have no current plans to quit) to reduce their smoking and eventually quit.

DETAILED DESCRIPTION:
Many smokers want to quit but have no plans to do so in the near future. Recent studies indicate that helping such smokers reduce the number of cigarettes they smoke each day, try medications to see that medications can help control their cravings, can make it easier for them to try to quit. This study tests whether a new medication (generic name = varenicline; brand name = Chantix) can help smokers in these ways.

The investigators will recruit 110 smokers in Vermont and 110 in Omaha, Nebraska, all of whom are interested in quitting some time in the future but have no current plans to quit. These smokers will be assigned by chance to receive either varenicline or a placebo. Neither the participants nor the scientists will know what the participants are receiving. Varenicline is a medication approved for smoking cessation in smokers who already have decided to quit. Varenicline both acts like nicotine to relieve craving and withdrawal when smokers try to quit and, importantly, also blocks the effects of nicotine from cigarettes. When smokers take varenicline and smoke, their cigarettes seem weaker and less beneficial. The investigators believe that making cigarettes less pleasing will make it easier for smokers to reduce, give them more control over their smoking, reduce their addiction to cigarettes, and make it easier for them to quit. After screening and giving consent, smokers will attend a first session to receive medication or placebo and to be instructed in how to use it to reduce their smoking. Smokers will be told they should use the medicine for at least 2 weeks and can use the medication for up to 2 months and, if they try to quit, they can receive an additional 3 months of medication after their quit date. Participants will be seen again at 2 weeks, 4 weeks and 2 months for brief help in reducing. After the first 2 months , they will be contacted by phone monthly for four more months. If participants are abstinent at 6 months they will be asked to return to provide a breath sample to verify abstinence. Participants will be asked to complete either written surveys or answer phone interviews and provide breath tests for which they will be reimbursed. The investigators will test, whether after 6 months, more smokers in the varenicline group tried to quit than in the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Able to get to research lab in Burlington, Vermont or Omaha, Nebraska
* Daily smoker
* Smoke at least 8 cigarettes per day
* No reduction in smoking in last 30 days
* No intention to quit in the next 30 days
* Never used Varenicline before
* Not currently using smoking cessation medications or nicotine replacement therapy
* Willing to use Varenicline for at least 2 weeks
* Fluent in English

Exclusion Criteria:

* Cannot be currently pregnant or breastfeeding
* Kidney disease
* Frequent nausea
* On certain medications for asthma and/or depression
* Another household member in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2008-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John R Hughes, MD, Principal Investigator — University of Vermont
Locations (2):
- United States (2):
  - Nebraska Medical Center, Omaha, Nebraska
  - University of Vermont, Burlington, Vermont

REFERENCES:
- [Result] Hughes JR, Rennard SI, Fingar JR, Talbot SK, Callas PW, Fagerstrom KO. Efficacy of varenicline to prompt quit attempts in smokers not currently trying to quit: a randomized placebo-controlled trial. Nicotine Tob Res. 2011 Oct;13(10):955-64. doi: 10.1093/ntr/ntr103. Epub 2011 Jun 7. PMID 21652735
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrolled sample size of 220; 2 were excluded because found to be ineligible after enrollment
Groups:
- Varenicline: 2 milligrams varenicline once per day for 2-8 weeks
- Placebo: Placebo once per day for 2-8 weeks
Period: Overall Study
Arm/Group | Varenicline | Placebo
Started | 107 | 111
Completed | 62 | 61
Not Completed | 45 | 50
Not completed — Lost to Follow-up | 45 | 50

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 107 | 111 | 218
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 99 | 106 | 205
  >=65 years | 8 | 5 | 13
Age Continuous [Mean (Standard Deviation); unit: years] | 44 (14) | 41 (15) | 42 (15)
Sex/Gender, Customized [Number; unit: participants]
  Female | 42 | 47 | 89
  Male | 64 | 63 | 127
  Missing | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 107 | 111 | 218

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Quit Attempt
Description: A quit attempt was defined as a self-reported attempt to quit smoking on a given day reported on a Time Line Follow Back (TLFB) obtained at each visit for the first 2 months and via monthly phone calls during months 3-6. The TLFB collected information for each day since the previous visit/call on number of cigarettes smoked that day, whether medication (varenicline or placebo) was used that day, and whether a quit attempt occured that day.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 107 | 111
participants | 55 | 36
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Test type: Superiority or Other; p = 0.06, Chi-squared; Odds Ratio (OR) = 1.7, 95% CI 2-sided [1.0 to 2.9]

2. Secondary Outcome: 7 Day Point Prevalent Abstinence Verified by Breath Carbon Monoxide of Less Than 10 Parts Per Million
Description: 7 day point prevalent abstinence 6 months after enrolling in the study was determined by two steps: (1) A report of no days of smoking for the 7 days prior to the 6 month on the Time Line Follow Back obtained at a telephone call 6 months after enrollment; (2) Those who reported no smoking for the prior 7 days came to our lab for breath carbon monoxide (CO) measurement to confirm abstinence. Breath CO had to be less than 10 parts per million for the participant to be classified as abstinent.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 107 | 111
participants | 15 | 8
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Test type: Superiority or Other; p = 0.10, Chi-squared; Odds Ratio (OR) = 2.1, 95% CI 2-sided [0.9 to 5.2]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) collected for 1 month after last dose of study medication, which varied from 2 weeks to 5 months
Description: Since this is a marketed drug we did not enter data about expected non-serious AEs into our database. The 0 non-serious AEs does not imply that no AEs were >5%, only that we did not capture that for analysis.
Arm/Group | Varenicline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/107 | 0/111
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No